CLINICAL TRIAL: NCT00144807
Title: Study of ACVBP Plus Rituximab in Previously Untreated Patients Aged From 18 to 59 Years With High Risk Diffuse Large B-cell Lymphoma (Age-adjusted IPI = 2-3)
Brief Title: ACVBP Plus Rituximab in Patients Aged From 18 to 59 Years With High-risk Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH03-3B
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Diffuse Large Cell Lymphoma
Keywords: lymphoma, diffuse large B-cell; rituximab; chemotherapy; autologous stem cell transplant
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-AC (Experimental): rituximab + doxorubicin + cyclophosphamide + autologous stem cell transplantation
  Interventions: Drug: rituximab; Drug: doxorubicin; Drug: cyclophosphamide; Procedure: autologous stem cell transplantation

INTERVENTIONS:
Drug: rituximab
Drug: doxorubicin
Drug: cyclophosphamide
Procedure: autologous stem cell transplantation

SUMMARY:
This study is a multicentric trial evaluating the efficacy of R-ACVBP in patients aged 18 to 59 years with high risk diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
This phase II non randomized study is based on the results of the LNH 98-5, LNH 87-2, LNH 93-3 and LNH 98-3B studies.

To date, the ACVBP regimen is considered as the reference induction treatment of the GELA in patients with 2-3 adverse prognostic factors. Indeed neither NCVBP regimen (LNH87-2) nor ECVBP (LNH93-3) led to increase the complete remission rate. More recently, the addition of etoposide to doxorubicin and cyclophosphamide (LNH98-3B) did not enhanced the complete remission rate with more toxicity. In patients < 60 years with 2-3 adverse prognostic factors the complete remission rate remained less than 65% in all these studies. Consequently, increasing the quality of response remains a major goal in this group of young patients with adverse prognostic factors.

It has been shown that the addition of rituximab to CHOP regimen significantly improved the CR rate in elderly patients with previously untreated large B-cell lymphoma when compared with CHOP alone without additional toxicities. Moreover, event-free survival and overall survival were found to be longer in the R-CHOP group. The present trial will evaluate the response rate obtained after four cycles of ACVBP combined to rituximab (R-ACVBP) before high dose therapy consolidative treatment in this group of higher risk patients.

The LNH87-2 study has shown that intensive consolidation treatment with autologous stem cell support was beneficial to high risk patients in good response after a full induction phase. The long-term results of this randomised study prompted us to consider high dose therapy as the best consolidative option for these patients.

ELIGIBILITY:
Inclusion Criteria:

Patient with histologically proven CD20+ diffuse large B-cell lymphoma (WHO classification).

Age from 18 to 59 years, eligible for transplant. Patient not previously treated. Age adjusted IPI = 2 or 3 With a minimum life expectancy of 3 months Negative HIV, HBV and HCV serologies < 4 weeks (except after vaccination). Having signed a written informed consent.

Exclusion Criteria:

Any history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in bone marrow or lymph node may be included.

Central nervous system or meningeal involvement by lymphoma. Contra-indication to any drug contained in the chemotherapy regimens. Poor renal function (creatinin level >150 mmol/l), poor hepatic function (total bilirubin level >30 mmol/l, transaminases >2.5 maximum normal level) unless these abnormalities are related to the lymphoma.

Poor bone marrow reserve as defined by neutrophils <1.5 G/l or platelets <100 G/l, unless related to bone marrow infiltration.

Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.

Any serious active disease (according to the investigator's decision). Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.

Pregnant or lactating women Adult patient under tutelage.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2003-12; Primary Completion 2008-09 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Complete remission rate (CR + CRu) | 12 weeks
  4 cycles of ACVBP

SECONDARY OUTCOMES:
Event-free survival and overall survival of patients submitted to autologous transplant and of the entire study population | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Fitoussi, MD, Principal Investigator — Lymphoma Study Association; Christian Gisselbrecht, MD, Study Director — Lymphoma Study Association; Corinne Haioun, MD, Study Chair — Lymphoma Study Association; Hervé Tilly, MD, Study Chair — Lymphoma Study Association
Locations (13):
- Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne, Belgium
- France (11):
  - Polyclinique Bordeaux Nord, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Hématologie CHU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital Saint Louis, Paris
  - Hématologie Adultes - Hôpital Necker, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Hématologie CHU Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif
- Schweirische Arbeitsgruppe fur klinische Krebsforschung, Lausanne, Switzerland

REFERENCES:
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Haioun C, Lepage E, Gisselbrecht C, Salles G, Coiffier B, Brice P, Bosly A, Morel P, Nouvel C, Tilly H, Lederlin P, Sebban C, Briere J, Gaulard P, Reyes F. Survival benefit of high-dose therapy in poor-risk aggressive non-Hodgkin's lymphoma: final analysis of the prospective LNH87-2 protocol--a groupe d'Etude des lymphomes de l'Adulte study. J Clin Oncol. 2000 Aug;18(16):3025-30. doi: 10.1200/JCO.2000.18.16.3025. PMID 10944137
- [Background] Tilly H, Lepage E, Coiffier B, Blanc M, Herbrecht R, Bosly A, Attal M, Fillet G, Guettier C, Molina TJ, Gisselbrecht C, Reyes F; Groupe d'Etude des Lymphomes de l'Adulte. Intensive conventional chemotherapy (ACVBP regimen) compared with standard CHOP for poor-prognosis aggressive non-Hodgkin lymphoma. Blood. 2003 Dec 15;102(13):4284-9. doi: 10.1182/blood-2003-02-0542. Epub 2003 Aug 14. PMID 12920037
- [Derived] Ghesquieres H, Larrabee BR, Haioun C, Link BK, Verney A, Slager SL, Ketterer N, Ansell SM, Delarue R, Maurer MJ, Fitoussi O, Habermann TM, Peyrade F, Dogan A, Molina TJ, Novak AJ, Tilly H, Cerhan JR, Salles G. FCGR3A/2A polymorphisms and diffuse large B-cell lymphoma outcome treated with immunochemotherapy: a meta-analysis on 1134 patients from two prospective cohorts. Hematol Oncol. 2017 Dec;35(4):447-455. doi: 10.1002/hon.2305. Epub 2016 Jun 10. PMID 27282998
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- [Derived] Fitoussi O, Belhadj K, Mounier N, Parrens M, Tilly H, Salles G, Feugier P, Ferme C, Ysebaert L, Gabarre J, Herbrecht R, Janvier M, Van Den Neste E, Morschhauser F, Casasnovas O, Ghesquieres H, Anglaret B, Brechignac S, Haioun C, Gisselbrecht C. Survival impact of rituximab combined with ACVBP and upfront consolidation autotransplantation in high-risk diffuse large B-cell lymphoma for GELA. Haematologica. 2011 Aug;96(8):1136-43. doi: 10.3324/haematol.2010.038109. Epub 2011 May 5. PMID 21546499
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org